CLINICAL TRIAL: NCT00490776
Title: A Phase II Study of Oral LBH589 in Adult Patients With Cutaneous T-Cell Lymphoma Who Are Intolerant to or Have Progressed on or After Prior HDAC Inhibitor
Brief Title: Study of Oral LBH589 in Adult Participants With Refractory/Resistant Cutaneous T-Cell Lymphoma (CTCL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was stopped on 15 June 2009 (early termination date) due to low prevalence of study population and slow accrual.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2212
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Cutaneous T-Cell Lymphoma
Keywords: Cutaneous T-Cell Lymphoma; adults; Mycosis Fungoides; Sézary Syndrome; CTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Panobinostat 20 mg (Experimental): Participants received panobinostat, 20 milligrams (mg), capsules, orally, thrice weekly on alternate Days 1, 3, and 5 per week of a 28-day treatment cycle until unacceptable toxicity, disease progression, and/or physician's discretion to discontinue the treatment.
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat — Panobinostat, 20 mg, hard gelatin capsules, orally, thrice weekly.
  Other Names: LBH589

SUMMARY:
This study evaluated the safety and efficacy of LBH589B in adult participants with refractory/resistant Cutaneous T-Cell Lymphoma and prior Histone Deacetylase (HDAC) inhibitor therapy.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent obtained prior to any screening procedures
2. Age greater than or equal to 18 years old
3. Participants with biopsy-confirmed stages IB-IVA mycosis fungoides or Sézary syndrome (SS). Participants with SS who have bone marrow involvement are also eligible. Participants with transformed CTCL are eligible
4. Participants must have been treated with an HDAC inhibitor given for the treatment of CTCL. Participants must have had disease progression on or following treatment with an HDAC inhibitor. Participants are also eligible if they had an inadequate response to an HDAC inhibitor defined as stable disease as the best response after at least 3 months of therapy. Participants previously treated with an HDAC inhibitor are also eligible if they experienced intolerance due to adverse events.
5. Baseline multiple-gated acquisition scan (MUGA) or echocardiogram must have demonstrated left ventricular ejection fraction (LVEF) ≥ the lower limit of the institutional normal
6. ECOG performance status ≤ 2

Exclusion criteria:

1. Participants with a history of visceral disease including central nervous system (CNS) involvement (i.e. stage IVB CTCL). Note, participants who have SS with bone marrow involvement are eligible
2. Impaired cardiac function
3. Concomitant use of drugs with a risk of causing torsades de pointes
4. Participants who have received chemotherapy or any investigational drug or undergone major surgery ≤ 3 weeks prior to starting study drug or who have not recovered from side effects of such therapy
5. Less than 3 months since prior electron beam therapy
6. Women who are pregnant or breast feeding, or women of childbearing potential (WOCBP) not willing to use a double method of contraception during the study and 3 months after the end of treatment.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-07-05 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2009-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- United States (18):
  - University of Alabama at Birmingham/ The Kirklin Clinic, Birmingham, Alabama
  - UCLA Medical Center School of Medicine/ Dpt of Hematology-Oncology, Los Angeles, California
  - University of Colorado Health Sciences Center/Anschutz Cancer Pavillion, Aurora, Colorado
  - Florida Academic Dermatology Centers, Miami, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Rush Presbyterian Hospital/St. Luke's Medical Center, Chicago, Illinois
  - St. Louis University Cancer Cennter, St Louis, Missouri
  - Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Clinical Cancer Center, New York, New York
  - Our Lady of Mercy Medical Center/Comprehensive Cancer Center, The Bronx, New York
  - Wake University Health Sciences, Winston-Salem, North Carolina
  - University of Oklahoma-Tulsa, Tulsa, Oklahoma
  - Craig Okada, Portland, Oregon
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - The Jones Clinic, Germantown, Tennessee
  - MD Anderson Cancer Center/University of Texas, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 9 participants were enrolled in the study at 8 investigative sites in the USA from 5 July 2007 to 15 June 2009. Recruitment was stopped on 15 June 2009 (early termination date) due to low prevalence of study population and slow accrual.
Groups:
- Panobinostat 20 mg: Participants received panobinostat, 20 mg, capsules, orally, thrice weekly on alternate Days 1, 3 and 5 per week of a 28-day treatment cycle until unacceptable toxicity, disease progression and/or physician's discretion to discontinue the treatment.
Period: Overall Study
Arm/Group | Panobinostat 20 mg
Started | 9
Completed | 0
Not Completed | 9
Not completed — Withdrawal by Subject | 1
Not completed — Administrative Problems | 1
Not completed — Death | 1
Not completed — New Cancer Therapy | 1
Not completed — Disease Progression | 5

BASELINE CHARACTERISTICS:
Population: Full Analyses Set (FAS) population was defined according to the Intention-to-Treat (ITT) principle and included all participants enrolled into the study.
Arm/Group | Panobinostat 20 mg
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) in Participants With Resistant Cutaneous T-Cell Lymphoma (CTCL) Treated With Oral Panobinostat by Using the Modified Severity-Weighted Assessment Tool (mSWAT)
Description: ORR was defined as the percentage of participants with best overall response (OR) of complete response (CR) or partial response (PR) based on mSWAT score, (OR = CR + PR). mSWAT score represents the product of the percentage total body surface area (%TBSA) involvement of each lesion type (patch, plaque, and tumor or ulceration), multiplied by a weighting factor: modified SWAT score = (patch %TBSA x 1) + (plaque %TBSA x 2) + (tumor or ulcer %TBSA x 4). The sum of these 3 numbers gave the modified SWAT score, on a 0 (no lesions) to 400 (lesions covering all areas) scale. CR based on mSWAT score was defined as the absence of skin disease. PR was defined as ≥ 50% decrease of the modified SWAT score compared to the Baseline score.
Time Frame: From first dose of study drug up to disease progression or death, (up to approximately 2 years)
Population: Since the study was terminated early due to low prevalence of study population and slow accrual Since the study was terminated early due to low accrual, no analyses were conducted for this study.
Arm/Group | Panobinostat 20 mg
Number analyzed (Participants) | 0

2. Secondary Outcome: Response Rate of Participants With Refractory CTCL Using the Physician's Global Assessment of Clinical Condition (PGA)
Description: Response rate was defined as the percentage of participants with CR or PR based on PGA scale. PGA is a 7-point grading scale for the investigator's assessment of the overall extent of improvement or worsening of the participant's disease as compared to Baseline. CR corresponds to Grade 0 (Completely clear) on PGA scale and was defined as no evidence of disease; 100% improvement. PR corresponds to Grade 2 (marked improvement) on PGA scale and was defined as significant improvement (≥75% - <90%); some evidence of disease remains.
Time Frame: From first dose of study drug up to disease progression or death, (up to approximately 2 years)
Population: as for outcome 1
Arm/Group | Panobinostat 20 mg
Number analyzed (Participants) | 0

3. Secondary Outcome: Response Rate in Participants With Refractory CTCL Using Modified Skin Score
Description: Response rate was defined as the percentage of participants with CR or PR based on mSWAT skin score. mSWAT score represents the product of the %TBSA involvement of each lesion type (patch, plaque, and tumor or ulceration), multiplied by a weighting factor: mSWAT score = (patch %TBSA x 1) + (plaque %TBSA x 2) + (tumor or ulcer %TBSA x 4). The sum of these 3 numbers gave the modified SWAT score, on a 0 (no lesions) to 400 (lesions covering all areas) scale. CR based on mSWAT score was defined as the absence of skin disease. PR was defined as ≥ 50% decrease of the modified SWAT score compared to the Baseline score.
Time Frame: From first dose of study drug up to disease progression or death, (up to approximately 2 years)
Population: as for outcome 1
Arm/Group | Panobinostat 20 mg
Number analyzed (Participants) | 0

4. Secondary Outcome: Responses in Index Lesions in Participants With Refractory CTCL by Lesion Measurements With Photographic Supporting Documentation
Description: Index lesions in each participant were selected as four to six of the prominent lesions amenable to bi-dimensional measurements. The longest diameter and its perpendicular measurement were used to determine the surface area and a weighted sum was determined as: Lesion 1 + lesion 2 + … + lesions 6 = Total sum of weighted score where Lesion 1: cm^2 x [1 (for patch); 2 (for plaque); 4 (for tumor or ulcer)]; Lesion 2: cm^2 x [1 (for patch); 2 (for plaque); 4 (for tumor or ulcer)]; Lesion 6: cm^2 x [1 (for patch); 2 (for plaque); 4 (for tumor or ulcer)]. These lesions were photographed at Baseline and at the time of response determined by either mSWAT or PGA
Time Frame: From first dose of study drug up to disease progression or death (up to approximately 2 years)
Population: as for outcome 1
Arm/Group | Panobinostat 20 mg
Number analyzed (Participants) | 0

5. Secondary Outcome: ORR of Participants With Resistant CTCL Treated With Oral Panobinostat by Using the Modified PGA to Assess Skin Disease and the Evaluation of Disease in the Viscera, Lymph Nodes and Blood (Circulating Sézary Syndrome Cells)
Description: ORR was defined as the percentage of participants with best OR of CR or PR based on PGA scale (OR = CR + PR). The PGA is a 7-point grading scale for the investigator's assessment of the overall extent of improvement or worsening of the participant's disease as compared to Baseline. CR corresponds to Grade 0 (completely clear) of PGA scale and was defined as no evidence of disease; 100% improvement. PR corresponds to Grade 2 (marked improvement) of PGA scale and was defined as significant improvement (≥75%-<90%); some evidence of disease remains.
Time Frame: From first dose of study drug up to disease progression or death, (up to approximately 2 years)
Population: as for outcome 1
Arm/Group | Panobinostat 20 mg
Number analyzed (Participants) | 0

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from first documented evidence of CR or PR until the earliest date of documented progression or death due to any cause among participants who achieved a confirmed CR or PR. The DOR was calculated in two ways. The DOR among responders only included participants who responded to the drug. The overall DOR included non-responders as having a DOR of zero days.
Time Frame: From first dose of study drug up to disease progression or death, (up to approximately 2 years)
Population: as for outcome 1
Arm/Group | Panobinostat 20 mg
Number analyzed (Participants) | 0

7. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as the time from the start of treatment until the first documented evidence of CR or PR among participants who achieved a confirmed CR or PR.
Time Frame: From first dose of study drug up to study completion (approximately 2 years)
Population: as for outcome 1
Arm/Group | Panobinostat 20 mg
Number analyzed (Participants) | 0

8. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the start of treatment until the earliest date of disease progression or death due to any cause, if sooner.
Time Frame: From first dose of study drug up to disease progression or death, (up to approximately 2 years)
Population: as for outcome 1
Arm/Group | Panobinostat 20 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event (AE): From the first dose of study drug up to 28 days after the last dose of study drug (up to approximately 2 years); Serious Adverse Event (SAE): From the first dose of study drug up to 4 weeks after the last dose of study drug (up to approximately 2 years)
Description: Safety population included all participants who received at least one dose of study drug and had at least one valid post-baseline assessment.
Arm/Group | Panobinostat 20 mg
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat 20 mg (N=9)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat 20 mg (N=9)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Sinus tachycardia (Cardiac disorders) | 1
Ear pruritus (Ear and labyrinth disorders) | 1
Dry eye (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 1
Fatigue (General disorders) | 4
Gait disturbance (General disorders) | 2
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 1
Pyrexia (General disorders) | 2
Thirst (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hordeolum (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Staphylococcal skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Postoperative fever (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Lymph node palpable (Investigations) | 1
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 1
Renal injury (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Lymphorrhoea (Vascular disorders) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to low accrual, no formal efficacy analyses were conducted for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.